CLINICAL TRIAL: NCT06014775
Title: A Prospective, One-arm and Open Clinical Study to Assess Safety and Efficacy of Anti-CD38 Antibody in the Treatment of Evans Syndrome
Brief Title: Anti-CD38 Antibody Treating Evans Syndrome
Acronym: 2023-D-ES
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023036
Record Dates: First submitted 2023-06-13; First posted 2023-08-28 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-10

CONDITIONS: Evan Syndrome; Treatment
MeSH Terms: conditions — Evans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention（Anti-CD38 antibody） (Experimental): 10 enrolled subjects : once a week x 8 doses
  Interventions: Drug: Anti-CD38 antibody Injection

INTERVENTIONS:
Drug: Anti-CD38 antibody Injection — intravenous Anti-CD38 antibody administration
  This study adopts a prospective, single arm, open design method. Ten subjects were enrolled in the study and were treated with Anti-CD38 antibody (16mg/kg/w) for 8 weeks.
  The first stage is the main research stage (d1-w8), which is the core treatment period. The subjects will receive intravenous infusion of 16mg/kg Anti-CD38 antibody once a week for 8 weeks to observe the safety and efficacy during treatment.
  The second stage (w9-w24) is the stage of withdrawal from the visit, mainly to observe the safety and continuous efficacy of Anti-CD38 antibody after treatment.

SUMMARY:
A single-center, open-label, off-label use investigator-initiated clinical study with safety run-in to explore the clinical activity and safety of Anti-CD38 Antibody in adult ES patients who have not responded adequately or relapsed after first-line treatment and at least one second-line therapy including immunosuppressive agents, Anti-CD20 Antibody and/or TPO-RA, or those in whom no other second-line treatment options are suitable.

DETAILED DESCRIPTION:
Evans' syndrome (ES) is defined as the concomitant or sequential association of warm auto-immune haemolytic anaemia (AIHA) with immune thrombocytopenia (ITP), and less frequently autoimmune neutropenia. ES is a rare situation that represents up to 7% of AIHA and around 2% of ITP. Due to the rarity of the disease, the treatment of ES is mostly extrapolated from what is recommended for isolated auto-immune cytopenia (AIC) and mostly relies on corticosteroids, rituximab, splenectomy, and supportive therapies.Despite continuous progress in the management of AIC and a gradual increase in ES survival, the mortality due to ES remains higher than the ones of isolated AIC, supporting the need for an improvement in ES management.

A branch of pathogenesis for ES has been revealed that plasma cells secrete pathogenic antibodies directed against platelet and red blood cell antigens. Antiplatelet specific plasma cells have been detected in the spleen of patients with rituximab refractory ITP. In those refractory cases, persistent autoreactive long-lived plasma cells in the bone marrow could explain treatment failure.

Anti-CD38 antibody, such as Daratumumab, has been developed to target tumoral plasma cells in multiple myeloma, was recently found to be effective in antibody-mediated diseases, such as autoimmune cytopenia following hematopoietic stem cell transplantation, systemic lupus and also ES.

This study will evaluate the safety and biologic activity of Anti-CD38 antibody in r/r primary ES who fail to respond to at least one previous second-line therapy or those who cannot chose suitable second-line therapy. The study will enroll approximately 10 participants. This trial will be conducted in China. All participants will be followed for at least 16 weeks after the 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 years.
* Prior to enrollment, a clinical diagnosis of primary Evans syndrome was made.
* Platelet count < 30×10^9/L or Hb < 100g/L or symptomatic anemia within 48 hours before the first administration of study drug;
* Failure to achieve response or relapse after corticosteroid therapy, and at least one second-line therapy or those who cannot chose other second-line therapy;
* If receiving emergency care for ES, treatment should be stopped >2 weeks before first dose.
* DAT positive (IgG+, with or without C3+).
* The patient need to be in the state of active hemolysis.
* With normal hepatic and renal functions.
* ECOG performance status ≤2.
* Cardiac function: New York Heart Association functional class ≤2.
* For patients receiving maintenance treatment, corticosteroids must have a stable dose at least 2 weeks before the first administration, TPO receptor agonists and azathioprine, danazol, cyclosporin A, tacrolimus, sirolimus, etc. must be stopped at least 4 weeks before the first administration; The end of anti-CD20 antibody treatment was>6 months.The end of alkylating agent treatment was>2 months.
* Understand the study procedures and voluntarily sign the informed consent form in person.

Exclusion Criteria:

* Secondary Evans syndrome. Received any treatment of anti-CD38 antibody drug
* Uncontrollable primary diseases of important organs, such as malignant tumors, liver failure, heart failure, renal failure and other diseases;
* HIV positive;
* Accompanied by uncontrollable active infection, including hepatitis B, hepatitis C, cytomegalovirus, EB virus and syphilis positive;
* Accompanied by extensive and severe bleeding, such as hemoptysis, upper gastrointestinal hemorrhage, intracranial hemorrhage, etc.;
* At present, there are heart diseases, arrhythmias that need treatment or hypertension that researchers judge is poorly controlled;
* Patients with thrombotic diseases such as pulmonary embolism, thrombosis and atherosclerosis;
* Those who have received allogeneic stem cell transplantation or organ transplantation in the past;
* Patients with mental disorders who cannot normally obtain informed consent and conduct trials and follow-up;
* Patients whose toxic symptoms caused by pre-trial treatment have not disappeared;
* Other serious diseases that may limit the subject's participation in this test (such as diabetes; Severe cardiac insufficiency; Myocardial obstruction or unstable arrhythmia or unstable angina pectoris in recent 6 months; Gastric ulcer, etc.);
* Patients with septicemia or other irregular severe bleeding;
* Patients taking antiplatelet drugs at the same time;
* Pregnant women, suspected pregnancies (positive pregnancy test for human chorionic gonadotropin in urine at screening) and lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of overall efficacy response after Anti-CD38 antibody treatment within 8 weeks | 8 weeks
  Overall response rate defined as improvement in any cytopenias by at least one grade, without worsening any other cytopenias or stable disease at least once within 8 weeks after the first dose.
Safety of Anti-CD38 antibody treatment | 24 weeks
  Incidence, severity, and relationship of treatment emergent adverse events after Anti-CD38 antibody treatment

SECONDARY OUTCOMES:
Evaluation of stable sustained response after Anti-CD38 antibody treatment at week 8 | 8 weeks
  Stable sustained response rate defined as improvement in any cytopenias by at least one grade, without worsening any other cytopenias or stable disease in 3 consecutive accessible assessments at least 7 days apart 8 weeks after the first dose.
Number of Participants With ES Response to Anti-CD38 antibody treatment | 24 weeks
  Complete response (CR) is complete resolution in all autoimmune cytopenias (neutropenia, anemia thrombocytopenia) maintained for more than two months, combined with an ability to wean off corticosteroids and/or other immunosuppressive medication. Partial response (PR) is improvement in any cytopenias by at least one grade, lasting more than two months, without worsening any other cytopenias or stable disease with the ability to wean corticosteroids and/or immunosuppressive medications by at least 50%. No response (NR) is no change in cytopenias with treatment, and the inability to wean corticosteroids or other immunosuppressive medications. Progressive disease (PD) refers to obtaining a CR or PR by the 3 month observation and relapsing or progressing by the 6 month observation, leading to cessation of study drug.
Measurements of platelet count at each visit time point | 24 weeks
  Platelet count at each visit time point
Measurements of Hb value at each visit time point | 24 weeks
  Hb value at each visit time point
Measurements of hemolytic marker reticulocyte count at each visit time point | 24 weeks
  hemolytic marker reticulocyte count at each visit time point
Measurements of hemolytic marker LDH at each visit time point | 24 weeks
  hemolytic marker LDH at each visit time point
Measurements of hemolytic marker haptoglobin at each visit time point | 24 weeks
  hemolytic marker haptoglobin at each visit time point
Measurements of hemolytic marker total bilirubin at each visit time point | 24 weeks
  hemolytic marker total bilirubin at each visit time point
Emergency treatment | 24 weeks
  Percentage of subjects who received emergency treatment
Duration of platelet response | 24 weeks
  The longest duration for which the subject sustained a platelet count ≥50×109/L and at least 2-fold from baseline at the meanwhile
Duration of Hb response | 24 weeks
  The longest duration for which the subject sustained a Hb level ≥100 g/L, or a Hb level increased more than 20g/L than baseline
Reduction of concomitant drug | 8 weeks
  Percentage of patients with reduced doses of corticosteroids and/or other concomitant immunosuppressive drugs at baseline by 8 weeks of treatment
Number of subjects with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale | 24 weeks
  Changes of the subjects' numbers in WHO bleeding score after Anti-CD38 antibody treatment according to the reported World Health Organization's Bleeding Scale. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Assessment of fatigue function in chronic disease treatment | 24 weeks
  The scores of Functional Assessment of Fatigue in Chronic Illness Therapy (FACIT-F) before and after Anti-CD38 antibody treatment
Health status survey | 24 weeks
  The change of Health status Questionnaire (SF-36) score before and after Anti-CD38 antibody treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, M.D, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months to 36 months after study completion
Access Criteria: Upon request to PI